CLINICAL TRIAL: NCT04252326
Title: The Knowledge, Attitudes and Practices of Healthcare Workers on Drug Hypersensitivity Reactions in Children: A Tertiary Center Experience
Brief Title: The Knowledge, Attitudes and Practices of Healthcare Workers on Drug Hypersensitivity Reactions in Children
Acronym: KAPHWDHRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nazlı ERCAN, Pediatric Allergy and Immunology Specialist, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: DrNazlı2020
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Adverse Drug Reactions
Keywords: Healthcare workers; Adverse drug reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Doctor (Active Comparator): Knowledge, Attitudes and Practices on Drug Hypersensitivity Reactions in Children
  Interventions: Other: Survey
- Nurse (Active Comparator): Knowledge, Attitudes and Practices on Drug Hypersensitivity Reactions in Children
  Interventions: Other: Survey
- Dentist (Active Comparator): Knowledge, Attitudes and Practices on Drug Hypersensitivity Reactions in Children
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Doctors, Nurses and Dentists filled survey about adverse drug reractions

SUMMARY:
Adverse drug reactions are an important public health consern that affects physician prescriptions and practice. The responsibilities of healthcare professionals in monitoring, prevention, treatment and reporting of drug hypersensitivity reactions and drug allergies are essential for patient safety. Providing drug safety must be one of the main goals to be achieved for every member of our society. In our study, we planned to evaluate the knowledge, attitudes, and behaviors of healthcare workers in our country about drug hypersensitivity reactions in pediatric patients and to determine the risk factors that may affect them.

DETAILED DESCRIPTION:
This study was carried out in a capital-located university hospital with a capacity of 1150 beds. Healthcare workers who are authorized to intervene in children (0-18 age group) including medical doctors, nurses and dentists were enrolled to study. In the evaluation of the knowledge, attitudes, and behaviors of the participants about drug hypersensitivity reactions in children, a study questionnaire was developed by pediatric allergy and immunology specialists and pediatric nurses by considering the other studies on the same subject.

ELIGIBILITY:
Inclusion Criteria:

The study included healthcare workers including medical doctors, nurses and dentists who perform interventions on children (0-18 years of age).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
we planned to evaluate the knowledge, attitudes, and behaviors of healthcare workers in our country about drug hypersensitivity reactions in pediatric patients | It is planned to fill the questionnaire in 2 hours.
  1. The knowledge level domain, consisted of 24 questions including mechanism of drug hypersensitivity reactions, clinical findings, diagnosis and treatment. The answer format was 3 options (yes/no /don't know). A triple variable scale was used for knowledge level (0 to 2: 0, false; 1, true; 2, do not know).
  2. The attitude domain consisted of 5 questions including the effect of DHRs on the patient's quality of life and advanced training and current diagnostic tests for the needs in this regard. A five-point Likert-type scale was used for the questions to determine the level of agreement or disagreement (1 to 5; 1 strongly disagree; 2, disagree; 3, uncertain; 4, agree; 5, strongly agree)
  3. The practice domain consisted of 9 questions including taking history and practice in drug allergy and advanced training in DHR. A Likert-type scale was used to determine the level of practices (1 - 5: 1, never; 2, very rarely; 3, sometimes; 4, often; 5, always).
we planned to evaluate the knowledge, attitudes, and behaviors of healthcare workers in our country about drug hypersensitivity reactions in pediatric patients | It is planned to fill the questionnaire in 2 hours.
  The knowledge level domain, consisted of 24 questions including mechanism of drug hypersensitivity reactions, clinical findings, diagnosis and treatment. The answer format was 3 options (yes/no /don't know).
  2. The attitude domain consisted of 5 questions including the effect of DHRs on the patient's quality of life and advanced training and current diagnostic tests for the needs in this regard. A five-point Likert-type scale was used for the questions to determine the level of agreement or disagreement The practice domain consisted of 9 questions including taking history and practice in drug allergy and advanced training in DHR. A Likert-type scale was used to determine the level of practices

SECONDARY OUTCOMES:
to determine the risk factors that may affect the knowledge, attitudes, and behaviors of healthcare workers in our country about drug hypersensitivity reactions in pediatric patient | It is planned to fill the questionnaire in 2 hours.
  Participants'demographic questions regarding the age, gender, profession, duration in the profession, title and educational status of the participants may effect their surveys scores

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Ercan, MD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Health Sciences University, Gülhane Training and Research Hospital, Gn. Dr. Tevfik Sağlam Cd No:11, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorji C, Tragulpiankit P, Riewpaiboon A, Tobgay T. Knowledge of Adverse Drug Reaction Reporting Among Healthcare Professionals in Bhutan: A Cross-Sectional Survey. Drug Saf. 2016 Dec;39(12):1239-1250. doi: 10.1007/s40264-016-0465-2. PMID 27743333
- [Result] Seid MA, Kasahun AE, Mante BM, Gebremariam SN. Healthcare professionals' knowledge, attitude and practice towards adverse drug reaction (ADR) reporting at the health center level in Ethiopia. Int J Clin Pharm. 2018 Aug;40(4):895-902. doi: 10.1007/s11096-018-0682-0. Epub 2018 Aug 9. PMID 30094559